CLINICAL TRIAL: NCT01593800
Title: The Effect of Probiotics on Lactose Intolerance
Acronym: PLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Ambrosia - SupHerb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PLI ver3
Record Dates: First submitted 2012-04-22; First posted 2012-05-08 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2012-02

CONDITIONS: Lactose Intolerance
Keywords: Probiotics; Lactose
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label probiotics (Experimental): Bio-25 is an innovative formula containing 11 different strains of unique probiotic bacteria and over 25 billion active bacteria in each capsule. All participants will receive either Probiotics (Bio-25,will be provided by SupHerb) or placebo pills blindly for six months. One day prior to each visit, subjects will be asked to consume lactose, fructose and sorbitol free foods, in order to avoid high base line of hydrogen from the presence of unabsorbed carbohydrates. Subjects will also be asked not to smoke 24 hours prior to each visit.
  Interventions: Dietary Supplement: Bio-25

INTERVENTIONS:
Dietary Supplement: Bio-25 — Bio-25 is an innovative formula containing 11 different strains of unique probiotic bacteria and over 25 billion active bacteria in each capsule. All participants will receive either Probiotics (Bio-25,will be provided by SupHerb) or placebo pills blindly for six months. One day prior to each visit, subjects will be asked to consume lactose, fructose and sorbitol free foods, in order to avoid high base line of hydrogen from the presence of unabsorbed carbohydrates. Subjects will also be asked not to smoke 24 hours prior to each visit.

SUMMARY:
Lactose intolerance (LI), also known as lactose malabsorption is the most common type of carbohydrate malabsorption. It is associated with the inability to digest lactose into its constituents, glucose and galactose, due to low levels of lactase enzyme activity (1-2). At birth, lactase activity is at the highest and it declines after weaning (1-2). The unabsorbed lactose is metabolized by colonic bacteria to produce gas (hydrogen (H2) and methane (CH4)) and short chain fatty acids. Symptoms related to LI appear 30 minutes to 2 hours after consumption of food products containing lactose. Related symptoms include: bloating, cramping, flatulence and loose stool (1-2, 17-18).

Highest rates of LI are found in the Asian populations, Native Americans and African Americans (60-100%), while lowest rates are found in people of northern European origin (including northern Americans) (3-4).

The diagnosis of LI based on patients' symptoms is sometimes problematic, since these symptoms are not specific and may differ from one patient to another. Breath hydrogen test have been advocated as the best diagnostic tool for the assessment of LI (15-16). During the test, subjects are sampled for hydrogen levels of breath samples at base line and every 30 minutes after the administration of 50 grams of oral lactose, for a total period of 180 minutes. A breath sample with > 20 ppm above baseline is considered positive for LI (15-16).

There are no established treatments for LI, other than almost complete avoidance of lactose rich dairy products. Avoidance of dairy products is a major concern since its outcome may result in a dietary calcium intake that is well below recommended dose of 1,000 mg per day for men and women and 1,300 mg for adolescents (8-10). For this reason different course of action needs to be considered instead of a complete exclusion of dairy products by LI patients.

Two possible interventions in the case of LI are the supplement of commercially available lactase (tablets) or the addition of probiotics.

The consumption of lactase enzyme as a food supplement may assist in restoring adequate levels of the enzyme needed for hydrolysis of lactose, especially for patients with low, or non existent levels of lactase. On the other hand, lactase products are problematic since not all lactase preparations are of the same concentration. Moreover, it is difficult to asses the amount of lactase tablets needed in order do fully hydrolyze lactose in each dairy mill (14).

Probiotics are live microorganisms that are commonly used in order to prevent or treat a disease. The current definition by the Food and Drug Administration and the World Health Organization is "Live microorganisms which, when administered in adequate amounts, confer a health benefit on the host." These microorganisms are a heterogeneous group, they are nonpathogenic and produce beta- galactosidase or lactase intracellularly that may assist in the digestion of lactose (11).

Studies have shown that people with lactose intolerance tolerated the lactose in yogurt better than the same amount of lactose in milk. The assumption was that the presence of lactase producing bacteria in the yogurt, especially Lactobacillus acidophilus, contributed to the digestion and absorption of lactose (5-6, 13).

It was also found that the presence of Lactobacillus bulgaricus and Streptococcus thermophilus alleviate lactose intolerance through their ability to produce lactase enzyme (7).

Finally, in another study it was found that consumption of milk containing Bifidobacterium longum resulted in significantly less hydrogen production and flatulence as compared to the consumption of control pasteurized milk (12).

Based on the mentioned data, the investigators speculate that the administration of probiotics may assist with the consumption of dairy products containing lactose. Therefore, the aim of this study is to evaluate the effect of probiotics on patients with LI.

DETAILED DESCRIPTION:
lactose hydrogen breath test (LHBT) will be performed at base line and at each visit (total of 7 breath samples from each patient). All subjects will be presented for the lactose hydrogen breath test after 8 hours fast.

At the initial stage, the subjects will take a base reading at time 0.

Subjects will then receive 50 g of lactose dissolved in a 100 ml of plain water and will perform further breath test samples every 30 minutes for 3 h. All breath samples will be end-expiratory and analyzed immediately by a Portable Breath Hydrogen Monitor (Gastro+ gastrolyzer, Bedfont Instruments, Holywell Lane, Upchurch, Kent, England). The concentration of breath hydrogen will be measured in parts per million (ppm). The measurements will then be plotted graphically and analyzed. The effect of probiotics on LI treatment will be measured by the following criteria:

1. If hydrogen levels measured after 6 months of treatment will be lower than levels measured at time 0 and/or patients will report a decrease of symptoms, the treatment of LI with Probiotics will be considered successful.
2. If hydrogen levels measured after 6 months of treatment will be the same or higher than levels measured at time 0 and/or patients will report an unchanged state or an increase of symptoms, the treatment of LI with probiotics will be considered unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* positive lactose hydrogen breath test (LHBT).

Exclusion Criteria:

1. Use of an antibiotic or Probiotics for more than 1 week before recruitment to the study
2. Use of lactase

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change of hydrogen levels measured due to probiotics administration | 2 years
  The effect of the probiotics on lactose intolerance will be evaluated through measurment of hydrogen levels (parts per million - ppm) at the end of each month of treatment. A decrease below cut off point of 20ppm will be considered as a successful outcome of the probiotics administration.

CONTACTS AND LOCATIONS:
Overall Officials: Tsachi T Perets, PhD, Study Director — Rabin Medical Center